CLINICAL TRIAL: NCT03706807
Title: Effect of the Mindfulness-Based Health Promotion Program - MBHP on Quality of Life and Maintenance of Cognitive Function in the Elderly: a Randomized Controlled Trial
Brief Title: Effect of the Mindfulness-Based Health Promotion Program (MBHP) in the Elderly: a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Mente Aberta de Mindfulness (Other)
Responsible Party: Principal Investigator, Marcelo Demarzo, MD, PhD, Principal Investigator, Centro Mente Aberta de Mindfulness
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 89700318.0.0000.5505
Record Dates: First submitted 2018-10-03; First posted 2018-10-16 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Quality of Life; Cognitive Impairment; Psychological
Keywords: Mindfulness; Older people; Quality of Life; Cognitive Function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Based Intervention (Experimental): This group will be included in the eight-week mindfulness program following the Mindfulness-Based Health Promotion (MBHP) protocol. The group will have a weekly meeting of an hour and thirty minutes for eight weeks to perform the mindfulness-based interventions accompanied by plus four one-hour meetings through a maintenance group after conclusion of the program, totaling 16 hours. The training will be lead by a certified instructor and he will introduce practices such as "mindfulness in breathing", "body scan", "mindful walking", "mindful movements" and "3-minutes of mindfulness" and the concepts of "first and second suffering" and the "Hi-Thanks-Bye".
  Interventions: Other: Mindfulness-Based Intervention
- Cognitive Stimulation (Active Comparator): The basic workshop is considered a cognitive stimulation and the participants will receive an hour and thirty minutes class once a week during four months. The abilities learned at the workshop will be basic computer functions from development of the psychomotricity involving the use of mouse, keyboard, MS paint, photo gallery and PowerPoint presentations to surf on the internet, learn how to play online games and use social networks. The activities of the workshop are elaborated according to the development of each class and is participants.
  Interventions: Other: Cognitive Stimulation
- Naïve (No Intervention): It's a waiting list group which will receive no intervention.

INTERVENTIONS:
Other: Mindfulness-Based Intervention — This intervention is a meditative practice which the individuals will practive in their daily life following the MBHP protocol
  Arms: Mindfulness-Based Intervention
Other: Cognitive Stimulation — A basic computer workshop in order to develop the psychomotricity involving the use of mouse, keyboard, MS paint, photo gallery and PowerPoint presentations to surf on the internet, learn how to play online games and use social networks
  Arms: Cognitive Stimulation

SUMMARY:
According to the World Health Organization (WHO), it is estimated that by 2025 the number of older people in Brazil will be approximately 33.4 million and it will be the sixth population in absolute numbers of the elderly in the world. The aging process is often associated with natural health debilitation, impairment of cognitive abilities, depression, loneliness and decreased daily life activity. Therefore, by increasing the number of older people also increase the needs and demands of health systems to serve this population. Government programs and projects that promote health and quality of life for this group must be developed and researched, so that the population aging happens in a satisfactory way and with physical and mental health. Several researches have been done on interventions that prevent the symptoms of memory impairment in elderly and on delaying symptoms of Mild Cognitive Impairment. Studies indicate that Mindfulness-Based Interventions (IBMs) are effective in the treatment of depression, anxiety, stress, chronic pain and in promoting well-being to young people and adults, yet the field of study of these interventions with the elderly is still a field to be explored and deepened. This project will focus on the discussion about the effectiveness of the Mindfulness-Based Health Promotion Program (MBHP) in the cognitive functions and quality of life of the elderly, based on quantitative and qualitative analysis. It will be used neuropsychological test and scales to assess the level of consciousness in the present moment, acceptance, self-compassion, quality of life and daily life activity, as well as a qualitative analysis through a structured script using the word evocation method and interviews through focus group.

DETAILED DESCRIPTION:
The MBHP-elderly study is a randomized and controlled trial of older people with 3 assessment point (baseline, post-intervention and six-months follow up) made with a cohort study whose participants will be older adults patients assisted in Primary Health Care of the Center for Aging Studies of the Federal University of São Paulo.

152 Participants will be recruited from the cohort and then randomized into the following groups: (I) MBHP intervention group (76 participants) in which the elderly will have a weekly meeting of an hour and thirty minutes for eight weeks to perform the mindfulness-based interventions accompanied by plus four one-hour meetings through a maintenance group after conclusion of the program, totaling 16 hours; (II) TAU control group (76 participants) of elderly who will take a cognitive simulation through computers for four months, a week meeting, totaling 16 hours. In both groups will be applied the same assessment for data collection and they will be applied in the baseline, post-intervention and six-month follow up. The steps of the study will be conducted based on Consolidated Standards of Reporting Trials (CONSORT) guidelines to report clinical studies in a clear, transparent and comprehensive manner. The protocol is reported according to the Standard Protocol Items: Recommendations for Intervention Trials (SPIRIT) statement.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 60 or over;
* be classified as cognitively normal or with mild cognitive impairment;
* know how to read and write.

Exclusion Criteria:

* practice contemplative practices such as yoga, reiki, tai-chi-chuan, vipassana, zen-buddhism, mindfulness and any other type of meditative practice in the last 6 months (with formal practice at least once / week);
* individuals with acute phase of depression;
* those with severe hearing or vision impairment;
* clinical diagnosis of schizophrenia or any other psychotic disorders;
* currently taking drugs that affect cognitive functions.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life-BREF (WHOQOL-BREF) | 51 months
  It was developed by the World Health Organization, the instrument is a short version of WHOQOL-100 and it comprises 26 items in which two are general about quality of life and the other 24 grouped into four domains related to quality of life and general health: physical health, psychological health, social relationships and environment. It presents Likert scale answer (1 to 5 points) and it is evaluated the mean of each subscale

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 51 months
  It assess the cognitive function. It is a 12-items test that measure eight cognitive domains: short-term memory (delayed drawing); visuospatial abilities (cube drawing, clock drawing); executive function (trail-making test; phonemic verbal fluency; verbal abstraction); attention, concentration, working memory; language; orientation to time. The test total score is 30 points where a score greater than or equal to 26 indicates normality and less than 25 points indicates Mild Cognitive Impairment.
Self-Compassion Scale | 51 months
  To measure the level of self-compassion of the individual. The Self-Compassion Scale consists of 26 items divided into 6 subscales for self-kindness; self-judgment; mindfulness; common humanity; and isolation. The answers are given in 5 points of the Likert scale which (1) is almost never and (5) is almost always.
Freiburg Mindfulness Inventory | 51 months
  it comprises 14 items that aim to identify through self-assessment the individual's perception of the frequency that the one experiences behaviors related to mindfulness (awareness to the present moment). The answers are marked on a Likert scale of 4 frequency levels: (1) Rarely; (2) Occasionally; (3) Fairly often; (4) Almost always. The total score ranges from 14 to 56 points and the higher the score the greater the mindfulness perception of the individual.
Depression Anxiety and Stress Scale - Short Form (DASS-21) | 51 months
  In order to assess psychological health we will use the DASS-21. It is a 21-item scale that measure and divide the symptoms of anxiety, depression and stress, in which participants indicate the degree to which they experienced these symptoms in the previous week on 7 items in each subscale: depression, anxiety and stress. It is a Likert-scale of 4 points between 0 to 3. The highest score in each subscale refer to more negative affective states.
Pittsburg Sleep Quality Index (PSQI) | 51 Months
  it is an instrument that evaluates the sleep quality of individual's the last month. It comprises 19 questions in self-report and 5 questions answered by some third party in which it will be made by phone call to a caregiver, relative or spouse. The components of the PSQI are C1 subjective sleep quality; C2 sleep latency; C3 sleep duration; C4 habitual sleep efficiency, C5 sleep disturbance, C6 Use of sleeping medication; C7 daytime dysfunction. Categorized as seven components in scores from zero (no difficulty) to three (severe difficulty). The sum of the results can range from zero to twenty-one scores, where the higher the number the worse quality of sleep.
The Duke University Religion Index | 51 months
  It is a 5-item scale that measure three major dimensions of religiousness: (1) organizational, the frequency of attending public religious activities and group-related; (2) nonorganizational, which involves religious activities performed in private, such as prayer, scripture study, watching religious TV or listening to religious radio; (3) Intrinsic religiosity, assessing the degree of personal religious commitment or motivations.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo MP Demarzo, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Centro Mente Aberta de Mindfulness e Promoção de Saúde, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided